CLINICAL TRIAL: NCT05041192
Title: The Effect of Synaquell on Objective Brain Function Measures in Ice Hockey Players
Brief Title: The Effects of Synaquell on Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: HealthTech Connex Inc. (Industry); Thorne HealthTech, Inc (Industry)
Responsible Party: Principal Investigator, Michael J. Stuart, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-004746
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: Ice Hockey; Cognitive Function; Cognition; Brain; Supplement; Contact Sport Athletes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synaquell Group (Experimental): Subjects will receive the dietary supplement, Synaquell, twice-daily during the hockey season.
  Interventions: Dietary Supplement: Synaquell
- Placebo Group (Placebo Comparator): Subjects will receive the placebo twice-daily, during the hockey season.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synaquell — 7.9 grams of Synaquell are mixed with 10 ounces of water two times per day. The daily amount taken by each participant is (15.8 grams).
  Arms: Synaquell Group
Dietary Supplement: Placebo — 7.9 grams of a placebo (that looks, smells, and tastes like Synaquell) are mixed with 10 ounces of water two times per day. The daily amount taken by each participant is (15.8 grams).
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to investigate the dietary supplement, Synaquell (TM), for effects on brain function.

DETAILED DESCRIPTION:
Ice Hockey players will be administered Synaquell over the course of one season. Each player will be administered Synaquell or a placebo twice, daily. They will be tested during the preseason and the postseason to compare changes in cognitive measures. This is an optimal population, as Synaquell was designed for contact sport athletes and others sustaining frequent head impacts.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater.
* Fluent English speakers.
* Medically cleared to play ice hockey.

Exclusion Criteria:

* An allergy to the ingredients of Synaquell or Synaquell+ (Magnesium, beta hydroxybutyrate, Glutathione, N-acetyl-L-cysteine, Riboflavin, Magnesium, Leucine, Isoleucine, Valine, Resveratrol, Curcumin Phytosome, Nicotinamide riboside, Docosahexanoic Acid).
* Clinically documented hearing issues.
* In-ear hearing aid or cochlear implant.
* Implanted pacemaker or defibrillator.
* Metal or plastic implants in skull.
* Lack of verbal fluency in the English language.
* History of seizures.
* Allergy to rubbing alcohol or EEG gel.
* Unhealthy scalp.

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Change in brain vital signs | Baseline, Postseason (approximately 6 months)
  Obtained by EEG recording of N100, P300, N400 amplitudes and latencies. Increased amplitudes are indicative of larger signals and increased latencies are indicative of slower responses.
Change in blood biomarker | Baseline, Postseason (approximately 6 months)
  Neurofilament light chain (NfL) blood serum levels.

SECONDARY OUTCOMES:
Change in King-Devick Test (KDT) scores | Baseline, Postseason (approximately 6 months)
  A rapid number-naming test that requires individuals to read 3 numbered cards a loud as fast as possible, the resulting time is the KDT score.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Stuart, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials